CLINICAL TRIAL: NCT02893761
Title: Bergonie Institute Breast Cancer Database
Status: Recruiting | Type: Observational
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Other Study IDs: IB BASE SEIN
Record Dates: First submitted 2016-08-18; First posted 2016-09-08 (Estimated); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: breast cancer; survival
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
A database of breast cancer patients was established at Institute Bergonié since the 90s , to assess patients' survival, assess practice, search for prognostic factors.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer
* Aged 18 years and over
* First treatment at Bergonie Institute

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with breast cancer treated at Bergonie Institute
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 1990-01 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2050-12 (Estimated)

PRIMARY OUTCOMES:
Distant metastasis-free survival at 5 years | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Gaetan Mac Grogan, MD, Principal Investigator — Institut Bergonié
Locations (1):
- Institut Bergonié, Comprehensive Cancer Center, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lhenaff M, Tunon de Lara C, Fournier M, Charitansky H, Brouste V, Mathoulin-Pelissier S, Pinsolles V, Rousvoal A, Bussieres E, Chassaigne F, Croce S, Ben Rejeb H, MacGrogan G. A single-center study on total mastectomy versus skin-sparing mastectomy in case of pure ductal carcinoma in situ of the breast. Eur J Surg Oncol. 2019 Jun;45(6):950-955. doi: 10.1016/j.ejso.2019.01.014. Epub 2019 Jan 17. PMID 30683448
- [Background] de Mascarel I, MacGrogan G, Debled M, Sierankowski G, Brouste V, Mathoulin-Pelissier S, Mauriac L. D2-40 in breast cancer: should we detect more vascular emboli? Mod Pathol. 2009 Feb;22(2):216-22. doi: 10.1038/modpathol.2008.151. Epub 2008 Sep 26. PMID 18820667
- [Background] de Mascarel I, Debled M, Brouste V, Mauriac L, Sierankowski G, Velasco V, Croce S, Chibon F, Boudeau J, Debant A, MacGrogan G. Comprehensive prognostic analysis in breast cancer integrating clinical, tumoral, micro-environmental and immunohistochemical criteria. Springerplus. 2015 Sep 21;4:528. doi: 10.1186/s40064-015-1297-8. eCollection 2015. PMID 26405647
- [Background] Ragage F, Debled M, MacGrogan G, Brouste V, Desrousseaux M, Soubeyran I, de Lara CT, Mauriac L, de Mascarel I. Is it useful to detect lymphovascular invasion in lymph node-positive patients with primary operable breast cancer? Cancer. 2010 Jul 1;116(13):3093-101. doi: 10.1002/cncr.25137. PMID 20564641
- [Background] Morgat C, MacGrogan G, Brouste V, Velasco V, Sevenet N, Bonnefoi H, Fernandez P, Debled M, Hindie E. Expression of Gastrin-Releasing Peptide Receptor in Breast Cancer and Its Association with Pathologic, Biologic, and Clinical Parameters: A Study of 1,432 Primary Tumors. J Nucl Med. 2017 Sep;58(9):1401-1407. doi: 10.2967/jnumed.116.188011. Epub 2017 Mar 9. PMID 28280221
- [Background] Mazroui Y, Mauguen A, Mathoulin-Pelissier S, MacGrogan G, Brouste V, Rondeau V. Time-varying coefficients in a multivariate frailty model: Application to breast cancer recurrences of several types and death. Lifetime Data Anal. 2016 Apr;22(2):191-215. doi: 10.1007/s10985-015-9327-y. Epub 2015 May 6. PMID 25944225
- [Background] Debled M, Auxepaules G, de Lara CT, Garbay D, Brouste V, Bussieres E, Mauriac L, MacGrogan G. Neoadjuvant endocrine treatment in breast cancer: analysis of daily practice in large cancer center to facilitate decision making. Am J Surg. 2014 Nov;208(5):756-763. doi: 10.1016/j.amjsurg.2013.12.032. Epub 2014 Apr 3. PMID 24814311
- [Background] Jones N, Gros A, Velasco V, Dapremont V, Brouste V, Gastaldello B, Debled M, Tunon de Lara C, Bonnet F, Barouk-Simonet E, Bubien V, Venat L, MacGrogan G, Longy M, Sevenet N. PTEN alterations in sporadic and BRCA1-associated triple negative breast carcinomas. Cancer Genet. 2022 Jun;264-265:8-15. doi: 10.1016/j.cancergen.2022.02.008. Epub 2022 Feb 25. PMID 35263698